CLINICAL TRIAL: NCT05233202
Title: Levosimendan Versus Placebo Before Tricuspid Valve Surgery in Patients With Right Ventricular Dysfunction
Acronym: LEONARD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200072
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-03

CONDITIONS: Patients Referred for an Isolated or a Combined Surgical Correction of Functional Moderate to Severe Tricuspid
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized (two arms, parallel groups); double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEVOSIMEDAN (Experimental): Levosimendan administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin 24H to 48H before anesthetic induction.
  Interventions: Drug: Levosimendan
- PLACEBO (Placebo Comparator): Placebo (isotonic sodium) administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin <48H before anesthetic induction.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Levosimendan — Levosimendan administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin 24H to 48H before anesthetic induction.
  Other Names: Experimental arm
  Arms: LEVOSIMEDAN
Drug: PLACEBO — Placebo (isotonic sodium) administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin <48H before anesthetic induction.
  Other Names: Control arm
  Arms: PLACEBO

SUMMARY:
A Prospective, multicenter, randomized (two arms, parallel groups); double-blind, placebo-controlled in order to assess the ability of preoperative levosimendan to prevent post-operative low cardiac output in high-risk patients referred to cardiac surgery for correcting functional tricuspid regurgitation. The primary end point is a composite element that includes peri-operative mortality and low cardiac output syndrome at day-90: 1) catecholamine infusion persisting beyond 48 hours after cardiac surgery, 2) the need for circulatory mechanical assist devices in the postoperative period, 3) or the need for renal replacement therapy at any time during intensive care unit stay. If a patient had at least 1 of these criteria, he or she was considered as meeting the primary end point.The secondary end points were 1) each component of the primary end point, and 2) the study drug safety defined as refractory hypotension.

DETAILED DESCRIPTION:
Patients referred for an isolated or a combined surgical correction of functional moderate to severe tricuspid are randomized in 2 arms, the levosimendan group or to the placebo group.

In the experimental group, levosimendan is administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin 24H to 48H before anesthetic induction.

In the comparator group, Placebo (isotonic sodium) administered as a continuous infusion over a 24-hour period at the rate of 0.2μg/kg/min, with no bolus administration. The infusion will begin <48H before anesthetic induction

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for an isolated or a combined surgical correction of functional moderate to severe tricuspid regurgitation [effective regurgitant orifice (ERO)>20mm², or systolic hepatic vein flow blunting or reversal]
* Written signed informed consent
* Affiliation to the French health care system (Sécurité Sociale)

Exclusion Criteria:

* Age < 18 years
* Severe organic renal dysfunction defined by creatinine clearance <30mL/min
* Recent endocarditis (<3 months)
* Recent myocardial infarction (<3 months)
* Tricuspid valve perforation or prolapse
* Cardiogenic shock requiring dobutamine support or cardiac assistance
* Severe liver injury (CHILD C)
* Left ventricular obstruction
* Allergy to levosimedan
* Current participation in other investigational drug or device studies or being in the exclusion period at the end of a previous study involving human participants, if applicable
* Pregnant or breastfeeding women
* Females of childbearing potential without effective method of birth control
* Patient on AME (state medical aid) unless exemption from affiliation
* Hypotension with SBP<90mmHg
* Severe tachycardia
* History of torsade de pointe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-01-23 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of CTAC on ventilation/perfusion ratios during a moderate to severe ARDS | day 90
  The primary end point is a composite element that includes peri-operative mortality and low cardiac output syndrome at day-90: 1) catecholamine infusion persisting beyond 48 hours after cardiac surgery, 2) the need for circulatory mechanical assist devices in the postoperative period, 3) or the need for renal replacement therapy at any time during intensive care unit stay. If a patient had at least 1 of these criteria, he or she was considered as meeting the primary end point.

SECONDARY OUTCOMES:
incidence of Refractory Hypotension (Drug safety) | day 90
  the study drug safety is defined as a refractory hypotension.
Number of catecholamine infusion | during 90 days
  persistence of infusion beyond 48 hours after cardiac surgery
Number of circulatory mechanical assist devices | during 90 days
  the need of circulatory mechanical assist devices in the postoperative period
Number of renal replacement therapy | during 90 days
  Need for renal replacement therapy at any time during intensive care unit stay

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris-Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No